CLINICAL TRIAL: NCT01388270
Title: The Effect of a Heparin-coated Dialysis Filter (Evodial) on Clotting and Intravascular Coagulation During Hemodialysis (HD) When Compared to a Conventional Polyflux Filter (170H)
Brief Title: Effect of a Pre Heparin Coated Dialysis Filter on Coagulation During Hemodialysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Solbjørg Sagedal, MD,PhD, Oslo University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2010/3019-2
Record Dates: First submitted 2011-06-29; First posted 2011-07-06 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Renal Failure
Keywords: Hemodialysis; Anticoagulation; Clotting; Coagulation; dalteparin; Clotting in the extracorporeal system during HD; Antithrombogenic property of Evodial HD filter; Anticoagulation during HD
MeSH Terms: conditions — Renal Insufficiency; Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Evodial (Active Comparator): a pre-heparin-coated hemodialysis filter
  Interventions: Device: a pre-heparin-coated hemodialysis filter; Hepran
- 170 H (No Intervention): Conventional filter

INTERVENTIONS:
Device: a pre-heparin-coated hemodialysis filter; Hepran — Use of the pre-heparin-coated filter compared to the conventional filter in a cross over design
  Other Names: HeprAN membrane; polyacrylonitrile; heparin-grafted membrane
  Arms: Evodial

SUMMARY:
The purpose of this study is to determine whether the heparin-coated dialysis filter is superior to a conventional filter during hemodialysis in twelve stable, chronic hemodialysis (HD) patients.

The antithrombogenic properties of the heparin-coated dialysis filter and of the conventional filter will be compared by means of statistical tests.

DETAILED DESCRIPTION:
In the present study twelve chronic hemodialysis (HD) patients will be included. Exclusion criteria are use of acetylsalicylic acid and/warfarin, clinical signs of infection and disseminated malignant disease. For each patient four HD sessions will be investigated; alternating with use of the pre-heparin-coated filter or the conventional filter. Dalteparin is reduced to 50% of the conventional dose and is given as one single bolus dose at start of HD.

The venous drip chamber will be visually inspected for evaluation of clot score during each HD session. The filter will be visually inspected for clot score at the end of each session.

Blood specimens will be drawn systematically during each HD session to evaluate platelet and coagulation activity as well as anti Factor Xa activity, haematology and urea/creatinine to evaluate dialysis effect.

The antithrombogenic properties of the pre-heparin-coated filter and the conventional filter will be compared by means of statistical tests. The hypothesis is that the pre-heparin-coated filter induces significantly less clot score in the extracorporeal system during hemodialysis and also significantly less intravascular activation of the coagulation system compared to the conventional filter.

ELIGIBILITY:
Inclusion Criteria:

* Stable HD patients of at least 18 years of age.
* HD treatment for at least one month.
* Dialysis time at least 4 hours three times per week.
* Stable Hemoglobin value of at least 11 g/dl during the last 4 weeks.

Exclusion Criteria:

* Use of warfarin and/or acetylsalicylic acid.
* Disseminated malignant disease.
* Clinical signs of infection.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-09; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Activation of the intravascular coagulation system during hemodialysis with use of a pre-heparin-coated filter compared to a conventional filter | Activation of the intravascular coagulation system is assessed during four dialysis sessions within a two weeks period for a single patient
  Blood specimens for analysis of prothrombin fragment 1+2 and beta-thromboglobulin will be drawn at start of hemodialysis and after three and four hours of all hemodialysis sessions.

SECONDARY OUTCOMES:
A secondary outcome measure is degree of clot score in the extracorporeal system during hemodialysis with use of a pre-heparin-coated filter compared to the conventional filter. | The degree of clot score in the extracorporeal system is assessed during four hemodialysis sessions that for a single patient take place within a time frame of two weeks
  Degree of clot score will be evaluated in the venous drip chamber as follows: 1=normal (no signs of clot). 2=fibrinous ring, 3=clot and 4=stop in dialysis due to high degree of clotting

CONTACTS AND LOCATIONS:
Overall Officials: Solbjørg Sagedal, PhD, Principal Investigator — Oslo University hospital, Ullevål
Locations (1):
- Department of nephrology, Oslo University Hospital, Ullevål, Oslo, Norway